CLINICAL TRIAL: NCT07359079
Title: A Prospective, Multicenter, Randomized, Parallel-Controlled, Subject-Blinded, Evaluator-Blinded, Non-Inferiority Clinical Trial to Evaluate the Efficacy and Safety of PEGDE-crosslinked Hyaluronic Acid Hydrogels for the Correction of Midface Volume Deficiency and/or Midface Contour Deficiency
Brief Title: The Correction of Midface Volume Deficiency and/or Midface Contour Deficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Jinsaixing Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-OM002-PCT01
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: the Correction of Midface Volume Deficiency and/or Midface Contour Deficiency

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject-Blinded, Evaluator-Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulate (Experimental)
  Interventions: Procedure: Stimulate
- Restylane Volyme (Active Comparator)
  Interventions: Biological: Restylane Volyme

INTERVENTIONS:
Procedure: Stimulate — the Correction of Midface Volume Deficiency and/or Midface Contour Deficiency
  Arms: Stimulate
Biological: Restylane Volyme — the Correction of Midface Volume Deficiency and/or Midface Contour Deficiency
  Arms: Restylane Volyme

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of PEGDE-crosslinked hyaluronic acid hydrogels for the correction of midface volume deficiency and/or midface contour deficiency, on the premise of ensuring the safety of the subjects and maintaining the scientific integrity of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 26 (including 26 years old), male or female;
* Subjects willing to correct midface volume deficiency and/or midface contour deficiency;
* According to the assessment by the blinded evaluators, subjects must have mild to severe midface volume deficiency and/or midface contour deficiency on each side (MMVS grade of 2 to 4). It is not required for both sides to have the same MMVS grade, but the difference in MMVS grade between the two sides must be ≤ 1 grade;
* Subjects are able to understand the objective of the study, voluntarily participate in the study and are willing to sign a written ICF.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will be ineligible for enrollment in the study:

  1. Subjects known to be allergic to hyaluronic acid products or to any component of the investigational medical device/control medical device; or subjects with a known history of severe allergies or anaphylactic shock.
* Subjects showing abnormal coagulation mechanism (activated partial thromboplastin time (APTT) >1.5 times the upper limit of normal) during the screening period, or those who have received any thrombolytic agent, anticoagulant or antiplatelet drugs (such as warfarin and aspirin) within 2 weeks before the screening.
* Having tattoos, piercings, prominent facial hair, keloids, deformities, non-healed wounds, abscesses, granuloma, malignancies or precancerous lesions, malignant tumors, or skin mass of unknown nature, etc. in the midface area that may affect the efficacy evaluation or increase the treatment risks.
* Judged by the investigators, subjects with active skin diseases, inflammation, or infections (such as herpes, eczema, acne, dermatitis, psoriasis, herpes zoster, fungal infections, papillomatosis, etc.) that may affect the assessment of midface.
* Subjects who have previously undergone facial surgery for wrinkle removal (such as subcutaneous separation and lifting, Superficial Musculo-Aponeurotic System (SMAS) separation and lifting, subperiosteal separation and combined wrinkle removal) or those intending to undergo facial surgery for wrinkle removal during the trial.
* Subjects who have previously undergone face surgical procedures (such as autologous fat grafting, absorbable catgut embedding treatment, liposuction, lipolysis, etc.) in the midface area, or those intending to undergo such treatments during the trial.
* Subjects who have previously undergone face surgical procedures (such as autologous fat grafting, absorbable catgut embedding treatment, liposuction, lipolysis, rhytidectomy, etc.) in other sites of face (except in the midface area) within 24 months prior to the screening period, or those intending to undergo such treatments during the trial.
* Subjects who have previously received any permanent filler treatments (such as polymethyl methacrylate, silicone, expanded polytetrafluoroethylene, etc.) or other unknown material injection therapy in the midface area, or those intending to undergo such treatments during the trial.
* Subjects who have received calcium hydroxylapatite, poly-L-lactic acid, poly-lactic acid, poly-di-spiralactic acid, polycaprolactone, etc. in the midface area within 24 months prior to the screening period, or those intending to undergo such treatments during the trial.
* Subjects who have received cross-linked hyaluronic acid injection in the midface area within 12 months prior to the screening period, or those intending to undergo such treatments during the trial.
* Subjects who have undergone any cosmetic treatments (such as botulinum toxin treatment, non-crosslinked sodium hyaluronate filler, collagen filler, radiofrequency treatment, focused ultrasound treatment, laser treatment, medium or deeper chemical peels, dermabrasion, photodynamic therapy or other ablation surgeries, etc. (except mesotherapy)) in the midface area within 6 months prior to the screening period, or those intending to undergo such treatments during the trial.
* Subjects who have received mesotherapy, photobiologic modulation therapy (red and blue light, etc., except laser therapy), intense pulsed light, microneedling (except radio frequency microneedles), very superficial or superficial chemical peels (such as retinol, alpha hydroxy acids, salicylic acid, etc.) in the midface area within 3 months prior to the screening period, or those intending to undergo such treatments during the trial.
* Subjects with active autoimmune diseases (such as inflammatory bowel disease) or a history of such diseases, as well as those with active connective tissue diseases (such as rheumatoid arthritis, scleroderma, and systemic lupus erythematosus) or a history of such diseases.
* Subjects who have received chemotherapy, immunosuppressive treatments, immunomodulators (such as monoclonal antibodies, etc.), or systemic corticosteroids (excluding inhaled corticosteroids) within 3 months prior to the screening period; or those who have received any drug treatments prior to screening that may affect efficacy evaluation or increase treatment risks in the investigator's judgment.
* Subjects with a history of keloids.
* Subjects with noticeable facial edema, as judged by the investigator, which may affect injection safety or effectiveness evaluation.
* Subjects with severe dysfunction of vital organs (brain, heart, lung, liver and kidney, etc.) based on evaluation by investigators, such as severe cardiovascular and cerebrovascular diseases (such as hospitalization for myocardial infarction or cardiac surgery within 3 months, a medical history of congestive heart failure or myocardial infarction, severe unstable arrhythmia, hypertrophic cardiomyopathy, severe aortic stenosis, aneurysm or stroke, etc.), severe lung diseases (such as moderate to severe pneumonia and respiratory failure, etc.), or uncontrolled diabetes mellitus, epilepsy, or history of severe mental illness, history of psychological illness, visual impairment, etc..
* Subjects with full dentures or any devices covering all or part of the upper palate, or with severe malocclusion, dental or maxillofacial deformities, or noticeable asymmetry around the mouth.
* Subjects who have undergone oral treatments (such as tooth extraction, orthodontics, or dental implants) within 3 months prior to the screening period that may affect efficacy evaluation, or those planning to undergo such treatments during the trial.
* Subjects planning to experience significant weight changes (weight change > 10%) during the clinical trial.
* Pregnant or breastfeeding female subjects, or subjects with plans for pregnancy during the clinical trial.
* Subjects who have participated or are participating in drug clinical trials within 3 months prior to the screening period, or who have participated or are participating in clinical trials for other medical devices within 1 month prior to the screening period (except those who have signed informed consent only and have not received any intervention).
* Other conditions that are considered by the investigator not suitable for enrollment in this study.

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
The effectiveness rate of improvement for midface volume deficiency and/or midface contour deficiency at 6 months after the last injection (as assessed by the blinded evaluators). | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Beijing, Beijing Municipality, China